CLINICAL TRIAL: NCT00691470
Title: A Randomized, Double Blind Comparison of ATI-5923, a Novel Vitamin K Antagonist, With Warfarin in Patients Requiring Chronic Anticoagulation
Brief Title: Comparison of ATI-5923, a Novel Vitamin K Antagonist, With Warfarin in Patients Requiring Chronic Anticoagulation
Acronym: EmbraceAC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ARYx Therapeutics (Industry)
Responsible Party: Daniel Canafax, ARYx Therapeutics, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLN-505
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2008-10

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Venous Thromboembolic Disease; Myocardial Infarction; Cardiomyopathy
Keywords: Anticoagulation; Vitamin K-dependent clotting factor inhibitor; Coumadin; Warfarin; Atrial fibrillation; Prosthetic heart valve; Venous thromboembolic disease; Myocardial infarction or cardiomyopathy; Patients with one or more of the following indications for chronic warfarin anticoagulation:; Atrial fibrillation (paroxysmal, persistent or permanent, not due to a reversible cause, documented by ECG) or atrial flutter;; A prosthetic heart valve in the aortic or mitral position that requires chronic anticoagulation;; A history of venous thromboembolic disease (DVT and/or PE) requiring long term anticoagulation (> 6 months);; A history of myocardial infarction or cardiomyopathy requiring anticoagulation.; Currently receiving chronic warfarin therapy for another indication not listed, with Sponsor approval.
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Myocardial Infarction; Cardiomyopathies | interventions — tecarfarin; Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. ATI-5923 (Experimental): Dose adjusted ATI-5923
  Interventions: Drug: ATI-5923
- 2. Coumadin (Active Comparator): Dose adjusted Coumadin (warfarin)
  Interventions: Drug: Coumadin (warfarin)

INTERVENTIONS:
Drug: ATI-5923 — Dose Adjusted based on INR.
  Arms: 1. ATI-5923
Drug: Coumadin (warfarin) — Dose adjusted based on INR.
  Arms: 2. Coumadin

SUMMARY:
The purpose of this research study is to test an experimental drug ATI-5923 vs Coumadin. The study is intended to demonstrate ATI-5923 is superior to Coumadin for keeping INR values in the desired therapeutic range. Patients who require chronic anticoagulation with one or more of the following conditions are eligible for the study: atrial fibrillation or atrial flutter, prosthetic heart valve, venous thromboembolic disease, or history of myocardial infarction or cardiomyopathy will be enrolled.

DETAILED DESCRIPTION:
The primary study objective is to evaluate whether ATI-5923 is superior to adjusted dose warfarin in the quality of anticoagulation as measured by interpolated INR time in therapeutic range. This is a Phase II/III multi-center, randomized, stratified, double blind, parallel group, active control study comparing ATI-5923 with Coumadin in patients who require chronic, oral anticoagulation. Up to 600 patients who successfully complete all screening assessments and meet all eligibility criteria will be enrolled in the study and receive study drug treatment for 6-12 months depending on time of study entry.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one or more of the following indications for chronic warfarin anticoagulation (the patient may either be a new candidate for anticoagulation or may already be receiving warfarin):

   1. Atrial fibrillation (paroxysmal, persistent or permanent, not due to a reversible cause, documented by ECG) or atrial flutter.
   2. A prosthetic heart valve in the aortic or mitral position that requires chronic anticoagulation.
   3. A history of venous thromboembolic disease (DVT and/or PE) requiring long term anticoagulation (> 6 months).
   4. A history of myocardial infarction or cardiomyopathy requiring anticoagulation.
   5. Currently receiving chronic warfarin therapy for another indication not listed, with Sponsor approval.
2. Male or female greater than 18 years of age.
3. Able and willing to sign IRB approved written informed consent to participate in the study.
4. Able and willing to follow instructions, to comply with protocol requirements, and to attend required study visits.

Exclusion Criteria:

1. Contraindications to anticoagulation as listed in the warfarin package insert (Appendix D), such as active bleeding or lesions at risk of bleeding such as gastric ulceration, colonic or cerebral AV malformations, cerebral or aortic aneurysms, pericarditis or endocarditis. Patients who have had recent (< 14 days from screening) surgery or invasive procedures or are about to undergo surgery or other invasive procedures, such as lumbar puncture. Patients with blood dyscrasias or inherited disorders of hemostasis. Patients with a history of hemorrhagic tendencies or prior serious hemorrhagic events such as hemorrhage within the cranium, eye, spinal cord, retroperitoneum, or gastrointestinal tract.
2. Laboratory evidence at screening of clinically significant active bleeding, such as unexplained positive occult blood in stool, or unexplained positive urinary blood that is more than trace positive for hemoglobin.
3. Concomitant use of other anticoagulant or antiplatelet agents that may add to the hemostatic burden such as clopidogrel, ticlopidine, heparin or low molecular weight heparin (LMWH), or regular use of non selective long acting NSAIDs that cannot be discontinued prior to initiating ATI 5923/warfarin dosing (daily use of 81-100 mg aspirin is allowed).
4. A life expectancy of < 1 year, end stage renal failure requiring dialysis, end stage pulmonary disease requiring home oxygen, severe heart failure (NYHA class IV).
5. Dementia, severe psychiatric disorder, or ongoing alcohol or substance abuse.
6. Laboratory screening values indicating severe anemia (Hb < 10 gm/L), thrombocytopenia (platelet count < 90,000/mcL), or active liver disease.
7. Patients with conditions that will interfere with determination of the INR using the INRatio device, i.e., hematocrit <30% or >55%. Patients with the antiphospholipid syndrome may have abnormal INR results and should not be enrolled.
8. History of non disabling ischemic stroke within the last 3 months, prior major disabling ischemic stroke, or any history of intracranial bleeding.
9. Pregnant or nursing women or women of childbearing potential who will not use adequate contraception, such as oral or implantable contraceptives, IUD, or barrier methods (IUD or condom) with spermicide.
10. Currently participating in another clinical trial at screening, treatment with an investigational drug within 30 days of the first dose of study medication, or patients who previously participated in an ATI-5923 trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Percent of time INR is in therapeutic range after the exclusion of the first 4 weeks of treatment, using the linear interpolation method of Rosendaal(Rosendaal, 1993). | After the first month through end of study.

SECONDARY OUTCOMES:
The proportion of all study recorded INR values that are within the target range, after the exclusion of the INR values from the first 4 weeks of treatment | After the first month through end of study
Proportion of time patients have significant deviations from therapeutic INR range. | After the first month through end of study
A composite of the following clinically important outcome events | After the first month through end of study

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Birmingham Heart Clinic, PC, Birmingham, Alabama
  - Cardiology PC, Birmingham, Alabama
  - The Heart Center, PC, Huntsville, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Southwest Heart, Tucson, Arizona
  - Escondido Cardiology Associates, Escondido, California
  - University of California San Diego Medical Center, San Diego, California
  - Progressive Clinical Research, Vista, California
  - New West Physicians Clinical Research, Golden, Colorado
  - Cardiology Associates of Fairfield County, PC, Norwalk, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Cardiology Associates of Fairfield County, PC, Trumbull, Connecticut
  - Florida Research Network, LLC, Gainesville, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Jacksonville Heart Center - Pavillon, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Heart Center - South, Jacksonville, Florida
  - St. Luke's Cardiology Associates, Jacksonville, Florida
  - Jacksonville Heart Center, Jacksonville Beach, Florida
  - Orlando Heart Center, Orlando, Florida
  - The Heart and Vascular Institute of Florida, Safety Harbor, Florida
  - Georgia Heart Specialists, Covington, Georgia
  - Northeast Georgia Heart Center, PC, Gainesville, Georgia
  - Fox Valley Clinical Research Center, LLC, Aurora, Illinois
  - Illinois Heart and Lung Research Center, Normal, Illinois
  - DuPage Medical Group, Winfield, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - McFarland Clinic PC, Ames, Iowa
  - Heart and Vascular Clinic, Lacombe, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Endeavor Medical Research, PLC, Alpena, Michigan
  - Steljes Cardiology, PC, Henderson, Nevada
  - Cardiovascular Research Institute, LLC, Canton, Ohio
  - Plaza Medical Group, PC, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Internal Medicine of Greer, Greer, South Carolina
  - Medical Associates Clinic, LLP, Pierre, South Dakota
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - York Clinical Research, Norfolk, Virginia
  - Daniel Gottlieb, MD, Burien, Washington

REFERENCES:
- See also: EmbraceAC Study Site — http://www.aryx.com/wt/page/ati5923